CLINICAL TRIAL: NCT05428566
Title: A Comparison of a Pulse-Based Diet and the Therapeutic Lifestyle Changes Diet on Reproductive and Metabolic Parameters in Women with Polycystic Ovary Syndrome
Brief Title: A Comparison of a PULSE Diet and the TLC Diet on Reproductive, Metabolic Parameters in Women with PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Collaborators: Abdul Hameed Shoman Foundation (Unknown)
Responsible Party: Principal Investigator, Shatha Hammad, Assistant Professor, Assistant Professor, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-2019/27
Record Dates: First submitted 2021-07-25; First posted 2022-06-23 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Polycystic Ovary Syndrome; Metabolic Syndrome
Keywords: Polycystic Ovary Syndrome; Metabolic Syndrome; Therapeutic Lifestyle Changes Diet; Pulse-Based Diet; Aerobic Exercise
MeSH Terms: conditions — Polycystic Ovary Syndrome; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulse-based diet (Experimental): The pulse diet will include two pulse-based meals; each pulse meal will be consisted of about one cup of non-oil seed pulses, different varieties of pulses (dried beans, peas, lentils, lupine, and chickpeas) will be used. Varieties of pulses will be included and the participants will be provided with recipes and preparation ideas, which would enhance the palatability of pulses, give different taste choices, and ease the follow of the prescribed diet and encourage the participants to consume it for the target duration.
  The diet is isocaloric and balanced with a fixed macronutrient composition of 28% fat, 55% carbohydrate, and 17% protein.
  Interventions: Dietary Supplement: Pulse-based diet
- TLC diet (Placebo Comparator): TLC group will be provided with instructions to follow the TLC guidelines and a sample diet plan will be individualized for each participant. The healthy TLC diet will be tailored for each participant according to their energy levels in order to achieve the following amount of nutrients: less than 7% of total calories of saturated fatty acids, up to 10% of total calories of polyunsaturated fat, up to 20% of total calories of monounsaturated fat, less than 200 mg a day of cholesterol, at least 5 to 10 grams a day of soluble fiber.
  The diet is isocaloric and balanced with a fixed macronutrient composition of 28% fat, 55% carbohydrate, and 17% protein.
  Interventions: Dietary Supplement: TLC diet

INTERVENTIONS:
Dietary Supplement: Pulse-based diet — An isocaloric, balanced diet with a fixed macronutrient composition of 28% fat, 55% carbohydrate, and 17% protein.
  The pulse diet will include two pulse-based meals; each pulse meal will be consisted of about one cup of non-oil seed pulses, different varieties of pulses (dried beans, peas, lentils, lupine and chickpeas) will be used.
  Arms: Pulse-based diet
Dietary Supplement: TLC diet — An isocaloric, balanced diet with a fixed macronutrient composition of 28% fat, 55% carbohydrate, and 17% protein.
  The healthy TLC diet will be tailored for each participant according to their energy levels in order to achieve the following amount of nutrients: less than 7% of total calories of saturated fatty acids, up to 10% of total calories of polyunsaturated fat, up to 20% of total calories of monounsaturated fat, less than 200 mg a day of cholesterol, at least 5 to 10 grams a day of soluble fiber.
  Arms: TLC diet

SUMMARY:
The main objective of the study is to evaluate the effectiveness of a lifestyle program for women with Polycystic Ovary Syndrome (PCOS). The investigators want to assess the efficacy of a pulse-based diet (i.e. a diet that contains lentils, chick-peas, and beans) on the clinical features, biochemical, and hormonal parameters of PCOS compared to the healthy therapeutic lifestyle changes diet.

DETAILED DESCRIPTION:
The main objective of the study is to identify the effect of pulses on a range of PCOS and metabolic syndrome features. In this parallel clinical trial, 110 (18-35 years old) women with PCOS will be recruited. Participants will be randomly assigned to either a pulse-based diet or a therapeutic lifestyle changes-based diet. The effect of a pulse-based diet on a range of reproductive and metabolic parameters will be evaluated. The results of this study are anticipated to evaluate the therapeutic merits of a pulse-based diet for women with PCOS which would influence dietary guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Diagnosis of PCOS in addition to insulin resistance (Homeostasis model assessment (HOMA)-insulin resistance index ≥ 2).
* Aged 18-35 years

Exclusion Criteria:

* Individuals that are Keto diet, vegetarian, pregnant, lactating, class 2 obese (body mass index (BMI) ≥35) current smoker, or if they have diabetes, cardiovascular, kidney, liver, or hormonal disease.
* Individuals taking any medication or supplementation known to affect lipid, glucose, or hormone levels, and/or body weight for at least the last 3 months.
* Any individual who has an allergy or intolerance to pulses.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 144 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Blood concentration of androgen hormone | Change from Baseline sample at 3 months
  Androgen hormone; testosterone will be evaluated for all participants across the 2 study arms
Ovarian volume | Change from Baseline ovarian morphology at 3 months
  An experienced ultrasonographer will evaluate the ovarian volume for each ovary.
Ovulatory dysfunction | During nine months
  Assessed by measuring the duration of the menstrual cycle
Lipid profile | Change from Baseline sample at 3 months
  Blood Cholesterol will be evaluated for all participants across the 2 study arms
Change in fat mass | Change from Baseline measurements at 3 months
  Body composition scan using InBody 120 (the body composition analyzer) will be evaluated for all participants across the 2 study arms
Physical activity | Change from Baseline point at 3 months
  The validated Arabic short form of the International Physical Activity Questionnaire (IPAQ) will be used to evaluate physical activity of all participants. And an overall total physical activity MET-minutes/week score can be computed as: Total physical activity MET-minutes/week = sum of Total (Walking + Moderate + Vigorous) MET- minutes/week scores.
  ( < 4 : Low), (4-6 Moderate) and ( >6: Vigorous)
Blood pressure | Change from Baseline Systolic Blood Pressure at 3 months
  In mmHg.(Systolic and Diastolic)

OTHER OUTCOMES:
Previous dietary consumption | Baseline point. (At the beginning of the study)
  A validated Arabic food frequency questionnaire will be completed by all participants to evaluate previous dietary consumption of these women and compare it with dietary recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: Shatha Hammad, PhD, Principal Investigator — The University of Jordan
Locations (2):
- Jordan (2):
  - The University of Jordan, Amman, Amman Governorate
  - Jordan University Hospital, Amman, Amman Governorate

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apridonidze T, Essah PA, Iuorno MJ, Nestler JE. Prevalence and characteristics of the metabolic syndrome in women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2005 Apr;90(4):1929-35. doi: 10.1210/jc.2004-1045. Epub 2004 Dec 28. PMID 15623819
- [Background] Asemi Z, Samimi M, Tabassi Z, Shakeri H, Sabihi SS, Esmaillzadeh A. Effects of DASH diet on lipid profiles and biomarkers of oxidative stress in overweight and obese women with polycystic ovary syndrome: a randomized clinical trial. Nutrition. 2014 Nov-Dec;30(11-12):1287-93. doi: 10.1016/j.nut.2014.03.008. Epub 2014 Mar 15. PMID 25194966
- [Background] Azziz R, Marin C, Hoq L, Badamgarav E, Song P. Health care-related economic burden of the polycystic ovary syndrome during the reproductive life span. J Clin Endocrinol Metab. 2005 Aug;90(8):4650-8. doi: 10.1210/jc.2005-0628. Epub 2005 Jun 8. PMID 15944216
- [Background] Baillargeon JP, Carpentier A. Role of insulin in the hyperandrogenemia of lean women with polycystic ovary syndrome and normal insulin sensitivity. Fertil Steril. 2007 Oct;88(4):886-93. doi: 10.1016/j.fertnstert.2006.12.055. Epub 2007 Jun 7. PMID 17559844
- [Background] Balen AH, Laven JS, Tan SL, Dewailly D. Ultrasound assessment of the polycystic ovary: international consensus definitions. Hum Reprod Update. 2003 Nov-Dec;9(6):505-14. doi: 10.1093/humupd/dmg044. PMID 14714587
- [Background] Barr S, Reeves S, Sharp K, Jeanes YM. An isocaloric low glycemic index diet improves insulin sensitivity in women with polycystic ovary syndrome. J Acad Nutr Diet. 2013 Nov;113(11):1523-1531. doi: 10.1016/j.jand.2013.06.347. Epub 2013 Aug 30. PMID 23999280
- [Background] Bhathena RK. Insulin resistance and the long-term consequences of polycystic ovary syndrome. J Obstet Gynaecol. 2011;31(2):105-10. doi: 10.3109/01443615.2010.539722. PMID 21281021
- [Background] Carmina E, Napoli N, Longo RA, Rini GB, Lobo RA. Metabolic syndrome in polycystic ovary syndrome (PCOS): lower prevalence in southern Italy than in the USA and the influence of criteria for the diagnosis of PCOS. Eur J Endocrinol. 2006 Jan;154(1):141-5. doi: 10.1530/eje.1.02058. PMID 16382003
- [Background] Chavarro JE, Rich-Edwards JW, Rosner BA, Willett WC. A prospective study of dietary carbohydrate quantity and quality in relation to risk of ovulatory infertility. Eur J Clin Nutr. 2009 Jan;63(1):78-86. doi: 10.1038/sj.ejcn.1602904. Epub 2007 Sep 19. PMID 17882137
- [Background] Corbould A. Effects of androgens on insulin action in women: is androgen excess a component of female metabolic syndrome? Diabetes Metab Res Rev. 2008 Oct;24(7):520-32. doi: 10.1002/dmrr.872. PMID 18615851
- [Background] den Besten G, van Eunen K, Groen AK, Venema K, Reijngoud DJ, Bakker BM. The role of short-chain fatty acids in the interplay between diet, gut microbiota, and host energy metabolism. J Lipid Res. 2013 Sep;54(9):2325-40. doi: 10.1194/jlr.R036012. Epub 2013 Jul 2. PMID 23821742
- [Background] Diamanti-Kandarakis E, Argyrakopoulou G, Economou F, Kandaraki E, Koutsilieris M. Defects in insulin signaling pathways in ovarian steroidogenesis and other tissues in polycystic ovary syndrome (PCOS). J Steroid Biochem Mol Biol. 2008 Apr;109(3-5):242-6. doi: 10.1016/j.jsbmb.2008.03.014. Epub 2008 Mar 12. PMID 18440223
- [Background] Douglas CC, Gower BA, Darnell BE, Ovalle F, Oster RA, Azziz R. Role of diet in the treatment of polycystic ovary syndrome. Fertil Steril. 2006 Mar;85(3):679-88. doi: 10.1016/j.fertnstert.2005.08.045. PMID 16500338
- [Background] Goss AM, Chandler-Laney PC, Ovalle F, Goree LL, Azziz R, Desmond RA, Wright Bates G, Gower BA. Effects of a eucaloric reduced-carbohydrate diet on body composition and fat distribution in women with PCOS. Metabolism. 2014 Oct;63(10):1257-64. doi: 10.1016/j.metabol.2014.07.007. Epub 2014 Jul 18. PMID 25125349
- [Background] Gower BA, Chandler-Laney PC, Ovalle F, Goree LL, Azziz R, Desmond RA, Granger WM, Goss AM, Bates GW. Favourable metabolic effects of a eucaloric lower-carbohydrate diet in women with PCOS. Clin Endocrinol (Oxf). 2013 Oct;79(4):550-7. doi: 10.1111/cen.12175. Epub 2013 May 20. PMID 23444983
- [Background] Graff SK, Mario FM, Alves BC, Spritzer PM. Dietary glycemic index is associated with less favorable anthropometric and metabolic profiles in polycystic ovary syndrome women with different phenotypes. Fertil Steril. 2013 Oct;100(4):1081-8. doi: 10.1016/j.fertnstert.2013.06.005. Epub 2013 Jul 2. PMID 23830153
- [Background] Ha V, Sievenpiper JL, de Souza RJ, Jayalath VH, Mirrahimi A, Agarwal A, Chiavaroli L, Mejia SB, Sacks FM, Di Buono M, Bernstein AM, Leiter LA, Kris-Etherton PM, Vuksan V, Bazinet RP, Josse RG, Beyene J, Kendall CW, Jenkins DJ. Effect of dietary pulse intake on established therapeutic lipid targets for cardiovascular risk reduction: a systematic review and meta-analysis of randomized controlled trials. CMAJ. 2014 May 13;186(8):E252-62. doi: 10.1503/cmaj.131727. Epub 2014 Apr 7. PMID 24710915
- [Background] Jayalath VH, de Souza RJ, Sievenpiper JL, Ha V, Chiavaroli L, Mirrahimi A, Di Buono M, Bernstein AM, Leiter LA, Kris-Etherton PM, Vuksan V, Beyene J, Kendall CW, Jenkins DJ. Effect of dietary pulses on blood pressure: a systematic review and meta-analysis of controlled feeding trials. Am J Hypertens. 2014 Jan;27(1):56-64. doi: 10.1093/ajh/hpt155. Epub 2013 Sep 7. PMID 24014659
- [Background] Karimzadeh MA, Javedani M. An assessment of lifestyle modification versus medical treatment with clomiphene citrate, metformin, and clomiphene citrate-metformin in patients with polycystic ovary syndrome. Fertil Steril. 2010 Jun;94(1):216-20. doi: 10.1016/j.fertnstert.2009.02.078. Epub 2009 May 21. PMID 19463994
- [Background] Katcher HI, Kunselman AR, Dmitrovic R, Demers LM, Gnatuk CL, Kris-Etherton PM, Legro RS. Comparison of hormonal and metabolic markers after a high-fat, Western meal versus a low-fat, high-fiber meal in women with polycystic ovary syndrome. Fertil Steril. 2009 Apr;91(4):1175-82. doi: 10.1016/j.fertnstert.2008.01.035. Epub 2008 Mar 10. PMID 18331737
- [Background] Kazemi M, McBreairty LE, Chizen DR, Pierson RA, Chilibeck PD, Zello GA. A Comparison of a Pulse-Based Diet and the Therapeutic Lifestyle Changes Diet in Combination with Exercise and Health Counselling on the Cardio-Metabolic Risk Profile in Women with Polycystic Ovary Syndrome: A Randomized Controlled Trial. Nutrients. 2018 Sep 30;10(10):1387. doi: 10.3390/nu10101387. PMID 30274344
- [Background] Luhovyy BL, Mollard RC, Panahi S, Nunez MF, Cho F, Anderson GH. Canned Navy Bean Consumption Reduces Metabolic Risk Factors Associated with Obesity. Can J Diet Pract Res. 2015 Mar;76(1):33-7. doi: 10.3148/cjdpr-2014-030. PMID 26067245
- [Background] Marinangeli CP, Jones PJ. Pulse grain consumption and obesity: effects on energy expenditure, substrate oxidation, body composition, fat deposition and satiety. Br J Nutr. 2012 Aug;108 Suppl 1:S46-51. doi: 10.1017/S0007114512000773. PMID 22916815
- [Background] Marsh KA, Steinbeck KS, Atkinson FS, Petocz P, Brand-Miller JC. Effect of a low glycemic index compared with a conventional healthy diet on polycystic ovary syndrome. Am J Clin Nutr. 2010 Jul;92(1):83-92. doi: 10.3945/ajcn.2010.29261. Epub 2010 May 19. PMID 20484445
- [Background] Mehrabani HH, Salehpour S, Amiri Z, Farahani SJ, Meyer BJ, Tahbaz F. Beneficial effects of a high-protein, low-glycemic-load hypocaloric diet in overweight and obese women with polycystic ovary syndrome: a randomized controlled intervention study. J Am Coll Nutr. 2012 Apr;31(2):117-25. doi: 10.1080/07315724.2012.10720017. PMID 22855917
- [Background] Moghetti P, Castello R, Negri C, Tosi F, Perrone F, Caputo M, Zanolin E, Muggeo M. Metformin effects on clinical features, endocrine and metabolic profiles, and insulin sensitivity in polycystic ovary syndrome: a randomized, double-blind, placebo-controlled 6-month trial, followed by open, long-term clinical evaluation. J Clin Endocrinol Metab. 2000 Jan;85(1):139-46. doi: 10.1210/jcem.85.1.6293. PMID 10634377
- [Background] Mollard RC, Luhovyy BL, Panahi S, Nunez M, Hanley A, Anderson GH. Regular consumption of pulses for 8 weeks reduces metabolic syndrome risk factors in overweight and obese adults. Br J Nutr. 2012 Aug;108 Suppl 1:S111-22. doi: 10.1017/S0007114512000712. PMID 22916807
- [Background] Moran LJ, Noakes M, Clifton PM, Tomlinson L, Galletly C, Norman RJ. Dietary composition in restoring reproductive and metabolic physiology in overweight women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2003 Feb;88(2):812-9. doi: 10.1210/jc.2002-020815. PMID 12574218
- [Background] Nybacka A, Carlstrom K, Stahle A, Nyren S, Hellstrom PM, Hirschberg AL. Randomized comparison of the influence of dietary management and/or physical exercise on ovarian function and metabolic parameters in overweight women with polycystic ovary syndrome. Fertil Steril. 2011 Dec;96(6):1508-13. doi: 10.1016/j.fertnstert.2011.09.006. Epub 2011 Sep 29. PMID 21962963
- [Background] Pittaway JK, Ahuja KD, Robertson IK, Ball MJ. Effects of a controlled diet supplemented with chickpeas on serum lipids, glucose tolerance, satiety and bowel function. J Am Coll Nutr. 2007 Aug;26(4):334-40. doi: 10.1080/07315724.2007.10719620. PMID 17906185
- [Background] Stamets K, Taylor DS, Kunselman A, Demers LM, Pelkman CL, Legro RS. A randomized trial of the effects of two types of short-term hypocaloric diets on weight loss in women with polycystic ovary syndrome. Fertil Steril. 2004 Mar;81(3):630-7. doi: 10.1016/j.fertnstert.2003.08.023. PMID 15037413
- [Background] Tayyem RF, Abu-Mweis SS, Bawadi HA, Agraib L, Bani-Hani K. Validation of a food frequency questionnaire to assess macronutrient and micronutrient intake among Jordanians. J Acad Nutr Diet. 2014 Jul;114(7):1046-1052. doi: 10.1016/j.jand.2013.08.019. Epub 2013 Nov 12. PMID 24231366
- [Background] Toscani MK, Mario FM, Radavelli-Bagatini S, Wiltgen D, Matos MC, Spritzer PM. Effect of high-protein or normal-protein diet on weight loss, body composition, hormone, and metabolic profile in southern Brazilian women with polycystic ovary syndrome: a randomized study. Gynecol Endocrinol. 2011 Nov;27(11):925-30. doi: 10.3109/09513590.2011.564686. Epub 2011 May 31. PMID 21627406
- [Background] Winham, D. M., & Hutchins, A. M. (2007). Baked bean consumption reduces serum cholesterol in hypercholesterolemic adults. Nutrition Research, 27(7), 380-386. Retrieved from http://www.sciencedirect.com/science/article/pii/S0271531707001066. doi:http://dx.doi.org/10.1016/j.nutres.2007.04.017
- [Background] Winham DM, Hutchins AM, Johnston CS. Pinto bean consumption reduces biomarkers for heart disease risk. J Am Coll Nutr. 2007 Jun;26(3):243-9. doi: 10.1080/07315724.2007.10719607. PMID 17634169
- See also: Campos-Vega R, Loarca-Piña G, Oomah BD. Minor components of pulses and their potential impact on human health. Food Research International. 2010;43:461-482 — https://doi.org/10.1016/j.foodres.2009.09.004